CLINICAL TRIAL: NCT05388474
Title: A Prospective and Retrospective Observational Study of Multidrug-Resistant Patient Outcomes With and Without Ibalizumab in a Real-World Setting: United States
Brief Title: A Prospective and Retrospective Observational Study of Multidrug-Resistant Patient Outcomes With and Without Ibalizumab
Acronym: PROMISE-US
Status: Active, not recruiting | Type: Observational
Sponsor: Theratechnologies (Industry)
Collaborators: Excelsus Statistics Inc. (Unknown); Health Psychology Research Group (HPR) (Unknown); ICON Clinical Research (Industry)
Responsible Party: Sponsor
Other Study IDs: TH-IBA-CTR-1003
Record Dates: First submitted 2022-04-01; First posted 2022-05-24 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections; Multi-Antiviral Resistance
Keywords: HIV; Drug resistance
MeSH Terms: conditions — HIV Infections | interventions — ibalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1 (No ibalizumab or Pre-ibalizumab treatment):: This cohort will be comprised of Heavily treatment-experienced (HTE) patients with Multi Drug Resistant (MDR) HIV who are not receiving ibalizumab. These patients will roll-over into cohort 2 if a change to their ARV regimen is made to include ibalizumab.
  Interventions: Other: No ibalizumab or Pre-ibalizumab treatment
- Cohort 2 (On ibalizumab treatment):: This cohort will be comprised of Heavily Treatment-Experienced patients (HTE) with Multi Drug Resistant (MDR) HIV who are starting treatment with an ARV regimen that includes ibalizumab. Patients already receiving ibalizumab prior to study entry may also be included in Cohort 2 if baseline viral load (VL) and cluster of differentiation 4 (CD4) count data are available prior to ibalizumab treatment. Recruited patients will be required to consent to provide their full retrospective ARV treatment and drug resistance history, as well as retrospective historical data from their medical records from 01 May 2018 to enrollment.
  Interventions: Biological: On ibalizumab treatment

INTERVENTIONS:
Other: No ibalizumab or Pre-ibalizumab treatment — Patient registry
  Other Names: Ibalizumab
  Groups: Cohort 1 (No ibalizumab or Pre-ibalizumab treatment):
Biological: On ibalizumab treatment — Patient registry
  Other Names: Ibalizumab
  Groups: Cohort 2 (On ibalizumab treatment):

SUMMARY:
The virological efficacy of ibalizumab has been clearly demonstrated in multiple clinical trials. This study will expand ibalizumab's clinical data set and allow a better understanding of the virologic response durability on ARV regimens with or without ibalizumab in a heterogeneous real-world patient population. Additional data on the efficacy and safety of ibalizumab and its impact on patient reported outcomes will be captured until study end.

Primary Objective:

To evaluate the long-term efficacy, safety, and durability of ibalizumab in combination with other ARVs by comparing the virologic, immunologic and clinical outcomes of patients receiving ibalizumab treatment versus patients not receiving ibalizumab.

Secondary Objective:

To assess the efficacy of ibalizumab in combination with other antiretrovirals by comparing the virologic, immunologic, clinical and patient reported outcomes of patients before and after they receive ibalizumab treatment.

To assess the long-term safety and tolerability of ibalizumab.

Other Objectives:

To assess risk factors/predictors of virologic and immunologic response. To assess efficacy and safety in special populations that enroll.

DETAILED DESCRIPTION:
Antiretroviral therapy (ART) for treatment of human immunodeficiency virus (HIV) has evolved tremendously over recent years. Newer medications have superior efficacy and tolerability, affording more convenient treatment regimens. The proportion of patients receiving antiretroviral (ARV) treatment that maintain viral suppression is approximately 85% in the United States. However, some patients may not be able to adhere to the prescribed ARV regimen or harbour strains of HIV that are resistant to most currently available therapies. Multi-drug resistant (MDR) HIV may be transmitted or result from incomplete viral suppression, which leads to accumulation of mutations in the viral genome over time. Patients with MDR HIV infection have significantly fewer available treatment options to construct a fully suppressive regimen. This ultimately results in shorter life expectancy, greater potential for transmission of MDR virus, increased morbidity and greater use of health resources. These comparisons are valid for the general population as well as people infected with non-MDR virus.

Ibalizumab, a humanized IgG4 monoclonal antibody that binds to a conformational epitope on domain 2 of the extracellular portion of the CD4 receptor, belongs to a new class of ARVs, CD4-directed post-attachment HIV-1 inhibitors, Ibalizumab exhibits no known cross-resistance with other ARV medications. Ibalizumab was approved by the FDA on March 6, 2018 and is indicated in combination with other ARVs for the treatment of HIV-1 infection in heavily treatment-experienced adults with MDR HIV-1 infection failing their current ARV regimen. It has been available commercially from April 2018.

The safety, efficacy and durability of response to ibalizumab treatment in combination with other ARVs have been demonstrated in clinical trials. This registry is designed to better understand the long-term efficacy and safety outcomes of MDR patients with and without ibalizumab in a real-world scenario.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is Heavily treatment-experienced (HTE), with limited treatment options and a history of treatment failure;
2. Based on recent or historical resistance assays and ARV history, patients must have documented Multi Drug Resistant (MDR) HIV-1 (e.g., laboratory report and documented past ARV treatment);
3. Received an appropriate HIV-1 resistance assay (genotypic or phenotypic testing) to devise an OBR (which may include an investigational ARV treatment) or will receive an appropriate resistance assay prior to initiating ibalizumab treatment;
4. Provide signed and dated informed consent to the Investigator, indicating that the patient (or, legally acceptable representative) has been informed of all pertinent aspects of the study, and is capable of understanding and willing to comply with the registry requirements. The consent will request to access the patient's medical, hospital, pharmacy, and vital statistics records as appropriate, as well as historical medical data for the full retrospective time period (01 May 2018 to enrollment). Further, consent will be provided for access to all available historical resistance and ARV treatment data;
5. ≥18 years of age or older at the time of screening;
6. Provide information on at least one alternate contact person of their choice (primary care physician, close relative or emergency contact) who can be contacted, should the patient be lost to follow-up over the course of the study;
7. Acknowledgement that in the event of their death, additional information can be obtained by contacting their primary care physician, a close relative, emergency contact or by consulting public or external databases (death registries, obituary listings) when available and verifiable. This is to be done in accordance with local regulatory requirements and laws;
8. Exceptionally, patients who may have started ibalizumab outside of the approved indication can also be included in Cohort 2 of the registry at the discretion of the investigator, provided they determine clinical utility.

Exclusion Criteria:

1. Pregnant or breastfeeding;
2. Unable to provide informed consent;
3. Hypersensitivity to ibalizumab or any of the excipients in ibalizumab;
4. Previous ibalizumab experience (Cohort 1 only)
5. Previously enrolled in Cohort 2 of this registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll Heavily treatment-experienced (HTE) adult patients infected with MDR HIV-1. For Cohort 2, the study will accept patients prescribed ibalizumab across study sites, including patients previously enrolled in Cohort 1 who subsequently initiated ibalizumab treatment. The decision to include ibalizumab in the treatment regimen will be clinical and independent of patient inclusion in the study.
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome measures | Maximum 36 months
  To compare the virologic, immunologic and clinical outcomes of patients receiving ibalizumab treatment vs. matched patients not receiving ibalizumab. And to evaluate the long-term efficacy and durability of ibalizumab in combination with other antiretrovirals. The following data will be collected:
  RELEVANT DISEASE AND PATIENT CHARACTERISTICS:
  * HIV Type
  * Duration of HIV infection
  * Gender
  * Age
  * Race/ethnicity
  * Vital signs (weight (kilograms), height (meters), systolic and diastolic blood pressure (mmHg))
  * Geographic location
  * AIDS-defining illnesses (CDC classification)
  * Comorbidities and other diagnoses
  * Concomitant medications
Primary Outcome measures | Maximum 36 months
  BASELINE DISEASE CHARACTERISTICS:
  * Pre-enrolment Viral Load (copies/ml)
  * Pre-enrolment CD4 count (cells/mm3)
  * Laboratory parameters: Hepatitis serology, CD4 (cells/mm3), CD8 (cells/mm3), HIV-RNA, HIV subtype
  * Historic Antiretroviral treatment (three years prior to enrolment)
  * Previous (three years prior to enrolment) and ongoing antiretroviral treatment
  * Genotypic and phenotypic resistance data and complete history
  * HIV subtype when available for patient
Primary Outcome measures | Maximum 36 months
  ON-TREATMENT INFORMATION:
  * CD4 count (cells/mm3)
  * Viral Load (copies/ml)
  * Weight (kilograms)
  * HIV subtype when available for patient
  * Concomitant medication review
  * Resistance testing review
  * Optimized Background Regimen review
  * New AIDS-Defining Events (CDC classification)
  * Adverse Reactions/Serious Adverse reactions review
  * Hospitalizations review
  * Ibalizumab discontinuation date and reason (e.g., lost to follow-up, death).

OTHER OUTCOMES:
Secondary Outcome measures | Maximum 36 months
  - Treatment satisfaction (associated with use of an ibalizumab-containing ARV regimen) will be assessed using the HIV Treatment Satisfaction Questionnaire status version (HIVTSQs12) at Ibalizumab day 0 treatment initiation (Day 0IBA) and at 6, 12 and 24 months following ibalizumab initiation for participants in cohort 2.
Secondary Outcome measures | Maximum 36 months
  - Change in treatment satisfaction (associated with the transition to an ibalizumab-containing ARV regimen) will be assessed using the HIV Treatment Satisfaction Questionnaire change version (HIVTSQc12) at 6 and 12 months after Day 0IBA for participants in cohort 2.
Secondary Outcome measures | Maximum 36 months
  - Adherence to Antiretroviral regimen, defined as the self-reported number of missed ARV doses in the prior week, will be assessed at Day 0IBA and at 6 and 12 months after Day 0IBA for all Cohort 2 patients starting ibalizumab treatment at the time of enrollment or transitioning from Cohort 1 to Cohort 2.
Secondary Outcome measures | Max 36 months
  - Cohort 2 patients will be asked whether they have had any difficulties with Ibalizumab IV infusions to evaluate the patient experience with IV administration.

CONTACTS AND LOCATIONS:
Overall Officials: Princy N Kumar, MD, Principal Investigator — Georgetown University
Locations (36):
- United States (36):
  - Ruane Clinical Research, Los Angeles, California
  - Mills Clinical Research, Los Angeles, California
  - BIOS Clinical Research, Palm Springs, California
  - UC San Diego Owen Clinic, San Diego, California
  - Yale University, New Haven, Connecticut
  - Circle Care Center, Stamford, Connecticut
  - Waterbury Hospital, Waterbury, Connecticut
  - Whitman Walker Health, Washington D.C., District of Columbia
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Aids Healthcare Foundation, Fort Lauderdale, Florida
  - Gary J. Richmond, M.D., PA, Fort Lauderdale, Florida
  - Midway Specialty Care Center Miami Beach, Miami Beach, Florida
  - Orlando Immunology Center (OIC), Orlando, Florida
  - Bliss Health, Orlando, Florida
  - Can Community Health, Tampa, Florida
  - St-Joseph's Comprehensive Research, Tampa, Florida
  - CAN Community Health, Tampa, Florida
  - Triple O Research Institute PA, West Palm Beach, Florida
  - Indiana University Health Inc., Bloomington, Indiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Las Vegas Research Center, Las Vegas, Nevada
  - I.D. Care Associates, PA, Hillsborough, New Jersey
  - Prime Healthcare Services - St Michael's Medical Center, Newark, New Jersey
  - SUNY Upstate Medical Center, Syracuse, New York
  - Amity Medical Group, Charlotte, North Carolina
  - The Roper St. Francis Ryan White Wellness Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prism Health North Texas, Dallas, Texas
  - North Texas Infectious Diseases Consultants, P.A, Dallas, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - UT Health Houston, Houston, Texas
  - St. Hope Foundation, Houston, Texas
  - Legacy Community Pharmacy Services, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Yearly interim analyses may be presented at scientific conferences and meetings.

REFERENCES:
- [Background] Armenia D, Di Carlo D, Flandre P, Bouba Y, Borghi V, Forbici F, Bertoli A, Gori C, Fabeni L, Gennari W, Pinnetti C, Mondi A, Cicalini S, Gagliardini R, Vergori A, Bellagamba R, Malagnino V, Montella F, Colafigli M, Latini A, Marocco R, Licthner M, Andreoni M, Mussini C, Ceccherini-Silberstein F, Antinori A, Perno CF, Santoro MM. HIV MDR is still a relevant issue despite its dramatic drop over the years. J Antimicrob Chemother. 2020 May 1;75(5):1301-1310. doi: 10.1093/jac/dkz554. PMID 31976521
- [Background] Burkly LC, Olson D, Shapiro R, Winkler G, Rosa JJ, Thomas DW, Williams C, Chisholm P. Inhibition of HIV infection by a novel CD4 domain 2-specific monoclonal antibody. Dissecting the basis for its inhibitory effect on HIV-induced cell fusion. J Immunol. 1992 Sep 1;149(5):1779-87. PMID 1380539
- [Background] Freeman MM, Seaman MS, Rits-Volloch S, Hong X, Kao CY, Ho DD, Chen B. Crystal structure of HIV-1 primary receptor CD4 in complex with a potent antiviral antibody. Structure. 2010 Dec 8;18(12):1632-41. doi: 10.1016/j.str.2010.09.017. PMID 21134642
- [Background] Gathe JC, Hardwicke RL, Garcia F, Weinheimer S, Lewis ST, Cash RB. Efficacy, Pharmacokinetics, and Safety Over 48 Weeks With Ibalizumab-Based Therapy in Treatment-Experienced Adults Infected With HIV-1: A Phase 2a Study. J Acquir Immune Defic Syndr. 2021 Apr 1;86(4):482-489. doi: 10.1097/QAI.0000000000002591. PMID 33427765
- [Background] Kilby JM, Eron JJ. Novel therapies based on mechanisms of HIV-1 cell entry. N Engl J Med. 2003 May 29;348(22):2228-38. doi: 10.1056/NEJMra022812. No abstract available. PMID 12773651
- [Background] Moore JP, Sattentau QJ, Klasse PJ, Burkly LC. A monoclonal antibody to CD4 domain 2 blocks soluble CD4-induced conformational changes in the envelope glycoproteins of human immunodeficiency virus type 1 (HIV-1) and HIV-1 infection of CD4+ cells. J Virol. 1992 Aug;66(8):4784-93. doi: 10.1128/JVI.66.8.4784-4793.1992. PMID 1378510
- [Background] Pearce N. Analysis of matched case-control studies. BMJ. 2016 Feb 25;352:i969. doi: 10.1136/bmj.i969. PMID 26916049
- [Background] Reimann KA, Burkly LC, Burrus B, Waite BC, Lord CI, Letvin NL. In vivo administration to rhesus monkeys of a CD4-specific monoclonal antibody capable of blocking AIDS virus replication. AIDS Res Hum Retroviruses. 1993 Mar;9(3):199-207. doi: 10.1089/aid.1993.9.199. PMID 8471310
- [Background] Reimann KA, Lin W, Bixler S, Browning B, Ehrenfels BN, Lucci J, Miatkowski K, Olson D, Parish TH, Rosa MD, Oleson FB, Hsu YM, Padlan EA, Letvin NL, Burkly LC. A humanized form of a CD4-specific monoclonal antibody exhibits decreased antigenicity and prolonged plasma half-life in rhesus monkeys while retaining its unique biological and antiviral properties. AIDS Res Hum Retroviruses. 1997 Jul 20;13(11):933-43. doi: 10.1089/aid.1997.13.933. PMID 9223409
- [Background] Raymond S, Piffaut M, Bigot J, Cazabat M, Montes B, Bertrand K, Martin-Blondel G, Izopet J, Delobel P. Sexual transmission of an extensively drug-resistant HIV-1 strain. Lancet HIV. 2020 Aug;7(8):e529-e530. doi: 10.1016/S2352-3018(20)30205-8. No abstract available. PMID 32763213
- [Background] Reimann KA, Khunkhun R, Lin W, Gordon W, Fung M. A humanized, nondepleting anti-CD4 antibody that blocks virus entry inhibits virus replication in rhesus monkeys chronically infected with simian immunodeficiency virus. AIDS Res Hum Retroviruses. 2002 Jul 20;18(11):747-55. doi: 10.1089/08892220260139486. PMID 12167266
- [Background] Sattentau QJ, Moore JP. The role of CD4 in HIV binding and entry. Philos Trans R Soc Lond B Biol Sci. 1993 Oct 29;342(1299):59-66. doi: 10.1098/rstb.1993.0136. PMID 7904348
- [Background] Song R, Franco D, Kao CY, Yu F, Huang Y, Ho DD. Epitope mapping of ibalizumab, a humanized anti-CD4 monoclonal antibody with anti-HIV-1 activity in infected patients. J Virol. 2010 Jul;84(14):6935-42. doi: 10.1128/JVI.00453-10. Epub 2010 May 12. PMID 20463063
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Zhang XQ, Sorensen M, Fung M, Schooley RT. Synergistic in vitro antiretroviral activity of a humanized monoclonal anti-CD4 antibody (TNX-355) and enfuvirtide (T-20). Antimicrob Agents Chemother. 2006 Jun;50(6):2231-3. doi: 10.1128/AAC.00761-05. PMID 16723592
- See also: EACS (2019). European Aids Clinical Society (EACS) Guidelines version 10. — http://www.eacsociety.org/guidelines/eacs-guidelines/eacs-guidelines.html
- See also: UNAIDS, 2019. Global AIDS Update 2019. Communities at the centre. Defending rights, breaking barriers, reaching people with HIV services — https://www.unaids.org/sites/default/files/media_asset/2019-global-AIDS-update_en.pdf